CLINICAL TRIAL: NCT03928951
Title: General Practitioner Reassessment of the Antibiotherapy of Urinary Infections Initially Treated in Emergency Departments
Brief Title: General Practitioner Reassessment of Urinary Infection Antibiotherapy Prescribed by Emergency Departments
Acronym: ATB-IU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-CHITS-01
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Urinary Tract Infections
Keywords: Urinary infections; Antibiotherapy; Emergency; Reassessment
MeSH Terms: conditions — Urinary Tract Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suffering from urinary infection: Patients consulting in one of Toulon - La Seyne sur Mer hospital emergency departments because of urinary infection
  Interventions: Other: General practitioner reassessment of urinary infection antibiotherapy prescribed by emergency departments

INTERVENTIONS:
Other: General practitioner reassessment of urinary infection antibiotherapy prescribed by emergency departments — Antibiotherapy will be prescribed by emergency physicians and general practitioners will be contacted 4 to 5 days later to know if antibiotherapy was modified

SUMMARY:
Urinary infections are at the origin of many emergency department consultations and antibiotic prescriptions. Increase of bacteria resistance to antibiotics is promoted by an inappropriate use of those antibiotics but initial prescription in emergency departments is complicated by brief clinical examinations, unavailable sampling results and risks of multi-resistant bacteria. Large diffusion of new recommendations for urinary infection management should improve the quality of initial antibiotic prescription. However emergency physicians have no knowledge of the reassessment of antibiotherapy 48 to 72 hours after initial prescription by general practitioners which is a quality criterion of good antibiotic use. The main purpose of this study is to estimate the reassessment rate by general practitioners of the urinary infection antibiotherapies prescribed in emergency departments. This will allow assessing the quality of initial antibiotic prescription and help to improve practices.

DETAILED DESCRIPTION:
Urinary infections are at the origin of many emergency department consultations and antibiotic prescriptions. Increase of bacteria resistance to antibiotics is promoted by an inappropriate use of those antibiotics but initial prescription in emergency departments is complicated by brief clinical examinations, unavailable sampling results and risks of multi-resistant bacteria. Large diffusion of new recommendations for urinary infection management should improve the quality of initial antibiotic prescription. However emergency physicians have no knowledge of the reassessment of antibiotherapy 48 to 72 hours after initial prescription by general practitioners which is a quality criterion of good antibiotic use. The main purpose of this study is to estimate the reassessment rate by general practitioners of the urinary infection antibiotherapies prescribed in emergency departments.

Patients will be informed during their consultation in one of Toulon - La Seyne sur Mer hospital emergency departments. If they don't express opposition to their data collection, they will be included. A form will then be completed by emergency physicians with initial prescribed antibiotherapy, patients' general practitioners contact information and if patients have a shared medical file or not. 4 to 5 days later, patients' general practitioners will be contacted to know if urinary analysis results were transferred from emergency department to practitioners, if antibiotherapy was modified and if patients' shared medical file was consulted.

ELIGIBILITY:
Inclusion Criteria:

* Every patient more than 18 years who was administered antibiotherapy for urinary infection in emergency department or for whom urinary infection was diagnosed in emergency department (cystitis, acute pyelonephritis, prostatitis)

Exclusion Criteria:

* Patients less than 18 years old
* Patients opposed to their data use
* Patients hospitalized more than 24 hours
* Patients taking antibiotherapy already before their arrival in emergency department
* Patients without sufficient reading capacities or understanding of french language to express opposition to their research participation
* Any other reason which, according to investigator, might interfere with research objective evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in emergency departments of Toulon La Seyne sur Mer hospital because of a urinary infection and to whom antibiotherapy is prescribed
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Rate of antibiotherapies modified by general practitioners | 6 months
  Number of antibiotic prescriptions modified by general practitioners divided by the total number of initial antibiotic prescriptions

SECONDARY OUTCOMES:
Rate of initial antibiotherapies not relevant to recommendations | 6 months
  Number of initial antibiotic prescriptions not relevant to recommendations divided by the total number of initial antibiotic prescriptions
Rate of initial antibiotherapies not consistent with recommendations | 6 months
  Number of initial antibiotic prescriptions not consistent (molecule, dose, period of time) with recommendations divided by the total number of initial antibiotic prescriptions
Rate of reassessments not relevant to recommendations | 6 months
  Number of antibiotic prescription modifications not relevant to recommendations divided by the total number of antibiotic prescription modifications
Rate of reassessments not consistent with recommendations | 6 months
  Number of antibiotic prescription modifications not consistent (molecule, dose, period of time) with recommendations divided by the total number of antibiotic prescription modifications
Frequence of use of shared medical file | 6 months
  Number of patients for which the shared medical file is used divided by the total number of patients enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Mouna EL OMRI, MD, Study Director — Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No